CLINICAL TRIAL: NCT04589104
Title: Expressive Writing for COVID-19 Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00105575
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Distress Due to COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expressive writing (Experimental): The expressive writing intervention consists of a 6-week, virtually-delivered writing program. Each week, participants meet for 90 minutes via Zoom and will be guided through writing prompts designed to encourage emotional expression and enhance personal resilience. The progression of writing exercises flows as follows:
  * Week 1: Writing to expressive difficult emotions
  * Week 2: Writing to release & integrate difficult emotions
  * Week 3: Writing to nurture gratitude
  * Week 4: Writing to enhance strengths & resources
  * Week 5: Writing to cultivate positive meaning & savor goodness
  * Week 6: Writing to invite insight, perspective, & growth
  Interventions: Behavioral: Expressive writing

INTERVENTIONS:
Behavioral: Expressive writing — The expressive writing intervention consists of a 6-week, virtually-delivered writing program. Each week, participants meet for 90 minutes via Zoom and will be guided through writing prompts designed to encourage emotional expression and enhance personal resilience. The progression of writing exercises flows as follows:
  * Week 1: Writing to expressive difficult emotions
  * Week 2: Writing to release & integrate difficult emotions
  * Week 3: Writing to nurture gratitude
  * Week 4: Writing to enhance strengths & resources
  * Week 5: Writing to cultivate positive meaning & savor goodness
  * Week 6: Writing to invite insight, perspective, & growth

SUMMARY:
The purpose of this study is to determine the impact of a 6-week, virtually-delivered expressive writing intervention on resilience in a cohort of individuals currently navigating the COVID-19 pandemic during spring 2020.

DETAILED DESCRIPTION:
The purpose of this study is to determine the impact of a 6-week, virtually-delivered expressive writing intervention on resilience in a cohort of individuals currently navigating the COVID-19 pandemic during spring 2020.

Eligible subjects will be adults who are able to read and write in English and are cognitively able to provide informed consent. Potential subjects will be recruited through the Duke Health & Well-Being email lists. The entirely virtual 6-week expressive writing intervention will be delivered via Zoom, REDCap, and email, and subjects will complete measures at baseline, 6 weeks, and 10 weeks (1 month post-intervention). Each week of the intervention will invite participants to complete a series of expressive writing assignments designed to support emotional expression and cultivate resilience, and the assignments will take approximately 60-90 minutes each week to complete.

The primary outcome is the 25-item Connor-Davidson Resilience Scale (CD-RISC). Other measures will include a basic demographics survey, questions about COVID-19 impact, post-writing surveys collected after the writing assignments, the 10-item Perceived Stress Scale (PSS), the Center for Epidemiologic Studies Depression Scale-Revised, and the 21-item Post -Traumatic Growth Inventory (PTGI). Participants will also have the option to share the content of their writing assignments with the research team if they choose.

The risks of participation in this study are minimal and include the risk of mild sadness after the writing assignments and the risk of loss of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects will be considered eligible if they feel they have been personally impacted by circumstances surrounding COVID-19. Other eligibility criteria include:

* Able to speak, read, write, and understand English
* Cognitively able to provide consent
* Ability to participate in a 6-week intervention delivered via Zoom, REDCap, and email

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Resilience | 3 months
  Connor-Davidson Resilience Scale (CD-RISC)

SECONDARY OUTCOMES:
Perceived stress | 3 months
  Perceived Stress Scale-10 (PSS10)
Depression symptoms | 3 months
  Center for Epidemiologic Studies Scale - Revised (CESDR)
Post-traumatic growth | 3 months
  Post Traumatic Growth Inventory (PTGI)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Glass, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Integrative Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bechard E, Evans J, Cho E, Lin Y, Kozhumam A, Jones J, Grob S, Glass O. Feasibility, acceptability, and potential effectiveness of an online expressive writing intervention for COVID-19 resilience. Complement Ther Clin Pract. 2021 Nov;45:101460. doi: 10.1016/j.ctcp.2021.101460. Epub 2021 Jul 27. PMID 34332289